CLINICAL TRIAL: NCT02814344
Title: Comparative Study of the Propagation of Uterine Electrical Activity (EHG) in Pregnant Women During Pregnancy and During Labour
Acronym: PropEHG
Status: Terminated | Type: Observational
Why Stopped: Investigator choice
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI10-PR-GONDRY
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Uterine Contraction; Pregnancy; Delivery, Obstetric
Keywords: labour

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- pregnant women not in labour: from 24 weeks of gestation until term, provided that they are not in labour
  Electrohysterography
  Interventions: Device: Electrohysterography
- women in labour: Electrohysterography
  Interventions: Device: Electrohysterography

INTERVENTIONS:
Device: Electrohysterography

SUMMARY:
The original aspect of the methodology proposed for this study concerns the use of as many as 16 electrodes to study the propagation and coordination (or synchronization) of uterine contraction. Over the last two years, the Compiègne University of Technology and the University of Reykjavik (Iceland) teams have developed the tools required to obtain good quality signals during electrohysterography and have worked on filtering and mapping of uterine electrical activity derived from these signals.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy

Exclusion Criteria:

* Minor patient
* twin pregnancy or more

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2011-08-09 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
parameter H2 | H2 value measured at each contraction during 1 hour
  To demonstrate a difference of propagation of the electrical signal during a physiological contraction of pregnancy and uterine contraction during delivery. The parameter H2 (nonlinear correlation coefficient) will be used to measure propagation of the electrical signal.

CONTACTS AND LOCATIONS:
Overall Officials: Jean GONDRY, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France